CLINICAL TRIAL: NCT01074541
Title: Vitamin D Production Depends on Ultraviolet-B Dose But Not on UV-intensity. A Randomized Controlled Trial
Brief Title: The Vitamin D Dose-Response Relationship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: The Danish Medical Research Council (Other)
Responsible Party: Morten Bogh MD, Bispebjerg Hospital, Department of Dermatology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 271-08-0461
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Vitamin D Status
Keywords: Vitamin D; UVB; Dose-Response; UV intensity; Skin cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Active Comparator): UV intensity 10 MIN
  Interventions: Radiation: UVB
- Group 2 (Active Comparator): UV intensity 5 MIN
  Interventions: Radiation: UVB
- Group 3 (Active Comparator): UV intensity 1 MIN
  Interventions: Radiation: UVB
- Group 4 (Active Comparator): UV intensity 20 MIN
  Interventions: Radiation: UVB

INTERVENTIONS:
Radiation: UVB — 0.375 SED x 4 in a week
  Other Names: UVB radiation
  Arms: Group 1; Group 2
Radiation: UVB — 0.75 SED x 4 in a week
  Other Names: UVB radiation
  Arms: Group 1; Group 2
Radiation: UVB — 1.5 SED x 4 in a week
  Other Names: UVB radiation
  Arms: Group 1; Group 2; Group 4
Radiation: UVB — 3.0 SED x 4 in a week
  Other Names: UVB radiation

SUMMARY:
The purpose of the study is to determine the importance of the UV intensity and the UVB dose on the Vitamin D response after UVB.

DETAILED DESCRIPTION:
The work is addressing vitamin D production after UVB exposure and explore the importance of UVB dose and UV intensity. Four different UVB doses and four different UV intensities are used to explore these relationships.

Many assumptions have been made concerning the vitamin D production after UVB exposure but only few studies exist.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* Healthy

Exclusion Criteria:

* Sun bed use
* Holiday or business travel south of 45 degrees latitude during trial
* Illness
* Drug addiction
* Pregnancy
* Lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Vitamin D (nmol/l) | 2 days after exposure
  Vitamin D measured in a blood sample to define the dose-response relationship between UVB dose, UV intensity and Vitamin D production in the skin after UVB exposure.

SECONDARY OUTCOMES:
Other parameters | 2 days after radiation
  To invesitage whether other parameters like sex, BMI, Diet etc. influences the vitamin D production after UVB exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Christian Wulf, Professor, Study Chair — Bispebjerg Hospital, Deparment of Dermatology
Locations (1):
- Bispebjerg Hospital, Department of Dermatology, Copenhagen NV, NV, Denmark